CLINICAL TRIAL: NCT01575028
Title: A Prospective, Double Blinded, Randomized Comparison of Transversus Abdominis Plane Block Versus Local Anesthetic Infiltration for Laparoscopic Appendectomy in the Pediatric Population
Brief Title: Transversus Abdominis Plane (TAP) Versus Local Anesthetic for Lap Appendectomies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was allowed to expire due to changes in standard care for the patient population within the NCH institution.
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Tarun Bhalla, MD, Assistant Clinical Professor, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB12-00140
Record Dates: First submitted 2012-04-05; First posted 2012-04-10 (Estimated); Results first posted 2015-06-01 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-07

CONDITIONS: Appendicitis
Keywords: Transversus abdominis plane block; TAP block; Local anesthetic infiltration; Appendectomy; Laparoscopic appendectomy
MeSH Terms: conditions — Appendicitis | interventions — Ropivacaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Local anesthetic infiltration injection (Active Comparator): Patients will receive local anesthetic infiltration injected at the surgical site by the surgeon at the end of surgery.
  Interventions: Drug: Bupivacaine
- Transversus abdominis plane (TAP) block (Experimental): Patients will receive a transversus abdominis plane (TAP) block.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — The TAP block will be delivered with 0.2ml/kg of 0.2% Ropivacaine with 1:200,000 epinephrine bilaterally
  Arms: Transversus abdominis plane (TAP) block
Drug: Bupivacaine — The local anesthetic at the incision sites will be injected by the surgeon.
  Arms: Local anesthetic infiltration injection

SUMMARY:
This study is a prospective, double-blinded, randomized comparison of 2 patient cohorts. One group of patients will receive a transversus abdominis plane (TAP) block. The second group will receive local anesthetic infiltration injected at the surgical site by the surgeon at the end of surgery for a laparoscopic appendectomy. The purpose of this study is to prospectively compare post-operative pain relief in pediatric patients undergoing laparoscopic appendectomy who have received either a transversus abdominis plane (TAP) block or local anesthetic infiltration by the surgeon for analgesia to compare the most appropriate delivery of effective analgesia. In an effort to improve postoperative analgesia while limiting opioid-related adverse effects, there continues to be an increased use of multimodal techniques in infants and children.

DETAILED DESCRIPTION:
The literature has clearly demonstrated that the effective treatment of postoperative pain in infants and children is challenging. Despite the recognition of the importance of postoperative analgesia and the potential adverse effects of postoperative pain, significant pain occurs during the postoperative period in both the inpatient and outpatients settings. Specifically, appendectomy is one of the most common pediatric surgical procedures and is associated with significant postoperative pain. Additionally, although the use of opioid analgesics is generally safe, adverse effects do occur thereby mandating the use of alternative analgesic techniques when feasible. In an effort to improve postoperative analgesia while limiting opioid-related adverse effects, there continues to be an increased use of multimodal techniques in infants and children. These can include TAP block as well as wound infiltration with local anesthetic. The efficacy of TAP blocks in the setting of laparoscopic appendectomy has been demonstrated in both adult and pediatric populations, however its efficacy in comparison to local anesthetic infiltration is unclear.

The TAP block was first described by McDonnell et al. in 2004 for pain control of procedures involving the anterior abdominal wall. The skin, muscles, and parietal peritoneum in this region are innervated by the T7 through L1 nerve roots. The authors described deposition of local anesthetic in the plane between the internal oblique and the transversus abdominis muscle where the terminal branches of the T7 through L1 nerves lie. Since then, the TAP block has been shown to effectively provide analgesia for a variety of abdominal procedures. In 2007 an ultrasound guided approach was described by Hebbard et al. with a subsequent study concluding that an ultrasound guided TAP block provided superior analgesia than a blind technique.

The frequency of surgical appendectomy in both the inpatient surgical as well as the ambulatory setting justifies this comparison of effective analgesia. This study can certainly change the daily practice of the pediatric anesthesiologist in providing optimal care in patient and family satisfaction, as well as recovery.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II
* Patients > 4 years of age
* Weight less than or equal to 60 kg
* Presenting for laparoscopic appendectomy

Exclusion Criteria:

* ASA physical status > II
* Patients < 4 years of age
* Weight greater than 60 kg
* Patients presenting for ruptured appendectomy surgical procedures
* Co-morbid diseases (cardiac, pulmonary (not including asthma), neurological disease)
* Patients having concomitant procedures (circumcision, orchiopexy, etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tarun Bhalla, MD, Principal Investigator — Nationwide Childrens
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] McDonnell JG, O'Donnell B, Curley G, Heffernan A, Power C, Laffey JG. The analgesic efficacy of transversus abdominis plane block after abdominal surgery: a prospective randomized controlled trial. Anesth Analg. 2007 Jan;104(1):193-7. doi: 10.1213/01.ane.0000250223.49963.0f. PMID 17179269
- [Background] Hebbard P, Fujiwara Y, Shibata Y, Royse C. Ultrasound-guided transversus abdominis plane (TAP) block. Anaesth Intensive Care. 2007 Aug;35(4):616-7. No abstract available. PMID 18020088

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Local Anesthetic Infiltration Injection | Transversus Abdominis Plane (TAP) Block
Started | 2 | 1
Completed | 2 | 0
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Local Anesthetic Infiltration Injection | Transversus Abdominis Plane (TAP) Block | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.425 (4.871965722) | 7.36 (0) | 11.40 (4.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Pain Relief
Description: Prospectively compare post-operative pain relief in pediatric patients undergoing laparoscopic appendectomy who have received either a transversus abdominis plane (TAP) block or local anesthetic infiltration by the surgeon for analgesia.
Time Frame: 12 hours post-operatively
Population: Due to changes in surgical technique & protocols by the general surgeons, we were only able to recruit 3 study subjects and the study was terminated. No analysis was performed.
Arm/Group | Local Anesthetic Infiltration Injection | Transversus Abdominis Plane (TAP) Block
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Local Anesthetic Infiltration Injection | Transversus Abdominis Plane (TAP) Block
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes